CLINICAL TRIAL: NCT01627626
Title: Effect of 0.1% Pilocarpine Mouthwash on Xerostomia : Double-blind, Randomized Controlled Trial
Brief Title: Effect of 0.1% Pilocarpine Mouthwash on Xerostomia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jeong-seong Kwon (Other)
Responsible Party: Sponsor-Investigator, Jeong-seong Kwon, Clinical assistant professor, Yonsei University
Organization: Yonsei University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 2-2011-0032
Record Dates: First submitted 2012-06-13; First posted 2012-06-26 (Estimated); Last update posted 2012-06-26 (Estimated); Status verified 2012-06

CONDITIONS: Xerostomia
Keywords: xerostomia; pilocarpine mouthwash; minor salivary gland secretion
MeSH Terms: conditions — Xerostomia | interventions — Pilocarpine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 0.1% pilocarpine mouthwash (Experimental): 0.1% pilocarpine solution which diluted 2% pilocarpine hydrochloride eyedrop with 0.9% saline
  Interventions: Drug: Pilocarpine
- 0.9% saline mouthwash (Placebo Comparator): 0.9% saline as a mouthwash
  Interventions: Drug: saline

INTERVENTIONS:
Drug: Pilocarpine — 0.1% pilocarpine solution which diluted 2% pilocarpine hydrochloride eyedrop with 0.9% saline.
  subjects were instructed to mouthwash with 10ml of solution for 1 minute.
  Arms: 0.1% pilocarpine mouthwash
Drug: saline — 0.9% saline solution
  Arms: 0.9% saline mouthwash

SUMMARY:
The aim of this study is to evaluate the effect of 0.1% pilocarpine mouthwash on subjective dryness, minor salivary flow rates and unstimulated whole salivary flow rate in xerostomic patients.

ELIGIBILITY:
Inclusion Criteria:

* xerostomia for 3 months or more, and
* adults aged 20 years and older.

Exclusion Criteria:

* acute asthma attack
* acute iritis
* narrow angle glaucoma
* pilocarpine allergy
* pregnancy
* lactating women, and
* person who was treating xerostomia with artificial saliva, pilocarpine, or etc.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2011-08; Primary Completion 2011-10 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Change from baseline in minor salivary flow rates at 60 minutes | before and after using the mouthwash (baseline, immediately, 30 minutes, 60 minutes)
  Minor salivary flow rates (from buccal, lower labial and palatal mucosa) were measured before and after using the mouthwash at predetermined times: baseline, immediately (0 min), and 30 and 60 minutes after. The Periotron 8000 device (Oraflow, New York, USA)was used to measure the flow rate (µl/cm2 per min) of saliva from the minor glands, in accordance with the method of Eliasson et al. (1996).

SECONDARY OUTCOMES:
Change from baseline in the severity of oral dryness at 60 minutes | Before and after using mouthwash (baseline, immediately, 30 minutes, 60 minutes)
  The severity of oral dryness was measured on a numerical rating scale (NRS ; 0-10, where 0=no dry mouth and 10=the worst dry mouth imaginable) before and after using the mouthwash at predetermined times: baseline, immediately (0 min), and 30 and 60 minutes after.
Change from baseline in the unstimulated whole salivary flow rates at 60 minutes | Before and after using mouthwash (baseline, 60 minutes)
  Unstimulated whole salivary flow rates (ml/min) were measured before and after using the mouthwash at predetermined times: baseline, and 60 minutes after. Unstimulated whole saliva was collected via the spitting method for 10 minutes while the subject was sitting in an upright position with the head slightly tilted forward and the eyes open after resting for 5 minutes. Subjects were instructed to minimize their orofacial movements during measurement.
Change from baseline in the severity of oral dryness, minor salivary flow rates, and the unstimulated whole saliva flow rate at 4 weeks | 4 weeks
  The severity of oral dryness, minor salivary flow rates, and the unstimulated whole salivary flow rates were measured after using the prescribed mouthwash regularly (with 10 ml of the solution for 1 minute, three times per day) for 4 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Jeong-Seung Kwon, DDS,MSD,PhD, Principal Investigator — Yonsei University Dental Hospital
Locations (1):
- Yonsei University Dental Hospital, Seoul, Seoul, South Korea